CLINICAL TRIAL: NCT02149537
Title: Risk Stratification for Clinical Severity of Sickle Cell Disease in Nigeria and Assessment of Efficacy and Safety During Treatment With Hydroxyurea
Brief Title: Risk Clinical Stratification of Sickle Cell Disease in Nigeria, Assessment of Efficacy/Safety of Hydroxyurea Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: University of Illinois at Chicago (Other); University of Ibadan (Other)
Responsible Party: Principal Investigator, Bamidele Tayo, Assistant profesor, Loyola University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205449
Record Dates: First submitted 2014-03-24; First posted 2014-05-29 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: sickle cell disease; sickle cell anemia; hydroxyurea; Nigeria; low income country; middle income country; developing country
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Adult patients to start to receive fixed low dose hydroxyurea (10 mg/kg) per day for six months and then crossover to no hydroxyurea treatment for six months, or start with no hydroxyurea treatment for six months and then crossover to receive fixed low dose hydroxyurea (10 mg/kg) per day for six months.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydroxyurea (Experimental): 500mg of hydroxyurea/day during 6 months
  Interventions: Drug: hydroxyurea
- No treatment (No Intervention): No hydroxyurea treatment during 6 months

INTERVENTIONS:
Drug: hydroxyurea
  Other Names: Hydroxycarbamide
  Arms: hydroxyurea

SUMMARY:
The vast majority of births with sickle cell disease (SCD) occur in Africa and 90% are thought to die before the age of five. Hydroxyurea (HU) is the only drug approved by the FDA for the treatment of sickle cell anemia. Although HU is used to treat small numbers of patients in Africa, cost, fear of toxicity, and lack of awareness and availability limit its use. The leukopenia that may be seen with HU raises the possibility of increased susceptibility to infection. Risk stratification - i.e., identification of patients most likely to benefit- could focus therapy and provide confidence that the risk:benefit ratio is favorable. Several clinical measures of future risk are well defined and findings on modifier genes in the US, primarily related to fetal hemoglobin (HbF), have further improved risk prediction. Whether the genetic variants predict severity in Africa is not known. The investigators have established a SCD cohort in Ibadan, Nigeria. In the first phase of this research the investigators will implement clinical risk examinations and assess the relationship between clinical characteristics (including levels of HbF) and known genetic markers. As a proxy for a birth cohort, the investigators will compare the frequency of the genetic markers in adult patients (i.e., "survivors") to children. In the second phase the investigators will randomize 40 high risk adult patients to fixed low dose HU or no HU treatment in a crossover design and monitor hematologic and physiologic parameters to document hematologic effects and safety. This work will lay the basis for a large-scale trial to document safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* HemoglobinSS (HbSS) or beta-zero (B0) thalassemia genotype
* Hemoglobin concentration >4.5 g/dL at steady state and time of enrollment
* Absolute neutrophil count >1,500/mircoliter
* Platelet count >95,000/microliter
* Serum creatinine <1.2 mg/dL
* Alanine transaminase less than two times the upper limit of normal

Exclusion Criteria:

* HIVpositive
* Hepatitis B and/or C positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Cytopenia | every 2 weeks during a period of 6 months
  Neutrophil count <500/microliter, platelet count <50,000 or a reticulocyte count<95,000 with Hemoglobin of 9.0 g/dL

SECONDARY OUTCOMES:
Development of infection evaluated by a physician at the point of care | every 2 weeks for period of 6 months
  Infections such as malaria or tuberculosis, which may be newly acquired or recrudescent.

OTHER OUTCOMES:
laboratory values of Hemoglobin F%, hemoglobin concentration, reticulocyte count, mean corpuscular volume and white blood cell count. | baseline, 3 months and 6 months.
Clinical complications such as acute pain episode, acute chest syndrome and need for blood transfusion. | every 2 weeks for a period of 6 months.
  Evaluated by a nurse or physician at point of care.

CONTACTS AND LOCATIONS:
Overall Officials: Bamidele O Tayo, PhD, Principal Investigator — Loyola University Chicago; Victor R Gordeuk, MD, Principal Investigator — University of Illinois at Chicago; Titilola S Akingbola, MBBS, FWACP, Principal Investigator — University of Ibadan College of Medicine, Nigeria; Richard S Cooper, MD, Principal Investigator — Loyola University Chicago; Lewis Hsu, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Ibadan College of Medicine, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saraf SL, Akingbola TS, Shah BN, Ezekekwu CA, Sonubi O, Zhang X, Hsu LL, Gladwin MT, Machado RF, Cooper RS, Gordeuk VR, Tayo BO. Associations of alpha-thalassemia and BCL11A with stroke in Nigerian, United States, and United Kingdom sickle cell anemia cohorts. Blood Adv. 2017 Apr 25;1(11):693-698. doi: 10.1182/bloodadvances.2017005231. PMID 28868518
- [Result] Tayo BO, Akingbola TS, Saraf SL, Shah BN, Ezekekwu CA, Sonubi O, Hsu LL, Cooper RS, Gordeuk VR. Fixed Low-Dose Hydroxyurea for the Treatment of Adults with Sickle Cell Anemia in Nigeria. Am J Hematol. 2018 May 14:10.1002/ajh.25143. doi: 10.1002/ajh.25143. Online ahead of print. No abstract available. PMID 29756251
- [Result] Akingbola TS, Tayo BO, Ezekekwu CA, Sonubi O, Zhang X, Saraf SL, Molokie R, Hsu LL, Han J, Cooper RS, Gordeuk VR. "Maximum tolerated dose" vs "fixed low-dose" hydroxyurea for treatment of adults with sickle cell anemia. Am J Hematol. 2019 Apr;94(4):E112-E115. doi: 10.1002/ajh.25412. Epub 2019 Feb 6. No abstract available. PMID 30663794
- Available data/document: Individual Participant Data Set: PR00007593 — http://doi.org/10.25934/PR00007593 — De-identified and anonymized IPD can be requested at http://doi.org/10.25934/PR00007593